CLINICAL TRIAL: NCT02358902
Title: Effect of Transcranial Direct Current Stimulation Associated With Aerobic Exercise Training for Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Nove de Julho (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08603612.0.0000.5511
Record Dates: First submitted 2014-12-19; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: Transcranial Direct Current Stimulation; Exercise; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): tDCS (tDCS - DC stimulator, Neurocom, Germany) / AE Group in which will receive active intervention of aerobic exercise training and active tDCS intervention
  Interventions: Device: tDCS; Procedure: active intervention of aerobic exercise
- Group B (Experimental): AE group which will receive active intervention of aerobic exercise and placebo tDCS (tDCS - DC stimulator, Neurocom, Germany)
  Interventions: Procedure: active intervention of aerobic exercise; Device: placebo tDCS
- Group C (Experimental): tDCS group which will receive placebo AE and active intervention for tDCS (tDCS - DC stimulator, Neurocom, Germany)
  Interventions: Device: tDCS; Procedure: placebo AE

INTERVENTIONS:
Device: tDCS — tDCS - DC stimulator, Neurocom, Germany
  Arms: Group A; Group C
Procedure: active intervention of aerobic exercise — different types of aerobic exercise
  Arms: Group A; Group B
Device: placebo tDCS — only 30 seconds of cortical stimulaion , with the power turned off for the remaining time (tDCS - DC stimulator, Neurocom, Germany)
  Arms: Group B
Procedure: placebo AE — the procedure was a training on the treadmill, but heart rate was maintained within 5% of the resting heart rate at the minimum speed on the treadmill
  Arms: Group C

SUMMARY:
This study consists of a randomized, double-blind, clinical trial with two months' duration of follow-up. The variable used was the VAS for pain, considering the values of any difference between the data before and after stimulation.

DETAILED DESCRIPTION:
The average between the analyzed values was 1.20, with a standard deviation of 0.84, taking into account a type I error of 5%, a type II error of 10% and a power of 80%. From the sample calculation was found an n = 10 for each group. The sample is amplified in order to avoid possible effects of dropout ending with a n = 15 in each group with a total N = 45.

Randomization was performed by a blinded therapist using sealed envelopes for each individual. The subjects will be divided into three intervention groups: tDCS (tDCS - DC stimulator, Neurocom, Germany) / AE Group, in which will receive active intervention of aerobic exercise training and active tDCS intervention. AE group, which will receive active intervention of aerobic exercise and placebo tDCS. And tDCS group, which will receive placebo AE and active intervention for tDCS.

Participants will be blinded to the intervention groups as well as therapists involved in the evaluation process.

The evaluation methods were carried out one week before the beginning of the intervention (baseline) for all variables. After the first week of intervention (neuromodulatory period) was performed ratings for level of cortical excitability (T1), and after the end of the one month period of intervention for all variables (T2). Follow-up evaluations were conducted one month (T3) and two months (T4) after the end of the intervention period."

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Fibromyalgia according to the American College of Rheumatology
2. Have completed high school
3. Age between 18 and 65 years old

Exclusion Criteria:

1. Were on medication for pain control for less than two months
2. In treatment of depression for less than two months
3. Patients with epilepsy, psychiatric disorders or who have any recent episode of neurologic disorders such as idiopathic syncope
4. Pregnant women and infants
5. Possessing metallic implant in the brain
6. In use of illicit drugs
7. That were in some kind of physical treatment for less than two months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Visual Numeric Scale (VNS) | Up to 2 months
  Pain intensity is measured using a scale from 0 to 10. A straight 10 cm line is displayed for the subject enumerated from zero to 10, where zero represents no pain and 10 the worst pain possible. Subjects should mark the number that most represents the symptom of pain at the moment. Outcome will be measured 24 hours after each intervention session, after 1 month of the end of protocol and 2 months after the end of protocol for evaluation of long term effects.

SECONDARY OUTCOMES:
Change in Visual Numeric Scale for Anxiety | Up to 2 months
  This scale has a straight 10 cm enumerated from zero to 10, where zero represents not anxious and 10 the most anxious possible. Subjects should mark the number that most represents the anxiety level at the moment. Outcome will be measured 24 hours after each intervention session, after 1 month of the end of protocol and 2 months after the end of protocol for evaluation of long term effects.

OTHER OUTCOMES:
Change in Pressure Pain Threshold (PPT) | Up to 2 months
  Using a pressure algometer (Wagner Instruments, USA), pressure is measured in the thenar region of the hand and at the uppermost portion of the anterior tibialis muscle. Pressure is held until the individual report onset of pain. At this time the amount of compression performed in kg/force is measured. Outcome will be measured after one week of intervention, after four weeks of intervention, after 1 month of the end of protocol and 2 months after the end of protocol, for evaluation of long term effects.
Change in Diffuse Noxious Inhibitory Control (DNIC-like effects) | Up to 2 months
  This parameter assesses through intense heterotopic stimulation, the response of endogenous pain modulation. Subjects emerge the hand in a container with ice-water (10-12˚C) for a period of one minute. During the last 30 seconds of immersion, the pressure pain threshold is measured in the other hand. The same procedure is performed for the other side. Temperature is measured by an immersion thermometer (ALLA BRAZIL 910.0150L). Outcome will be measured after four weeks of intervention, after 1 month of the end of protocol and 2 months after the end of protocol, for evaluation of long term effects.
Change in SF-36 questionnaire of quality of life | Up to 2 months
  This questionnaire evaluates different aspects in individual life such as: Vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Through different questions a score is generated for each subscale where zero represents the worst quality of life and 100 the best quality of life. Outcome will be measured after four weeks of intervention, after 1 month of the end of protocol and 2 months after the end of protocol, for evaluation of long term effects.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Simis, MD PhD, Study Chair — Institute of Physical Medicine and Rehabilitation, Clinicas Hospital, Faculty of Medicine, University of Sao Paulo

REFERENCES:
- [Result] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529